CLINICAL TRIAL: NCT02753465
Title: A Prospective Randomized Clinical Study for Laparoscopic D3 Lymph Node Dissection With Preservation of Left Colic Artery in Rectal Cancer Surgery
Brief Title: A Prospective Clinical Study for Laparoscopic D3 Dissection With Preservation of Left Colic Artery in Rectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, LI XIN-XIANG, professor of colorectal surger, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUDANLCA
Record Dates: First submitted 2016-04-03; First posted 2016-04-27 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Rectal Neoplasms
Keywords: Rectal Neoplasms; anastomosis; OS; DFS; LCA; laparoscopic surgery
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- left colic artery group (Experimental): Laparoscopic D3 Lymph Node Dissection with preservation of the left colic artery
  Interventions: Procedure: left colic artery
- High ligation group (Active Comparator): Laparoscopic D3 Lymph Node Dissection with high ligation
  Interventions: Procedure: High ligation

INTERVENTIONS:
Procedure: left colic artery — Laparoscopic D3 Lymph Node Dissection with preservation of left colic artery
  Arms: left colic artery group
Procedure: High ligation — Laparoscopic D3 Lymph Node Dissection with ligation above the left colic artery
  Arms: High ligation group

SUMMARY:
During surgery for rectal cancer, there is considerable controversy regarding the optimal level of ligation of the inferior mesenteric artery. Several studies have demonstrated the benefit of high ligation of the inferior mesenteric artery for the rectal cancer in order to achieve block dissection of lymph node metastases along the root of the inferior mesenteric artery. In contrast, other studies have shown a significant decrease in blood flow after inferior mesenteric artery clamping that may increase the risk of anastomotic ischemia and the long-term outcomes were not significantly different between high ligation of the inferior mesenteric artery and low ligation. So, a modified procedure was suggested to dissect fatty tissues and nodes in the angle between the inferior mesenteric artery and the left colic artery and the artery was ligated below the left colic artery. In the present clinical trial, the investigators perform laparoscopic surgery with this management strategy in rectal cancer. Thus, the goal of this study is to investigate the short-term and oncologic long-term outcomes associated with laparoscopic lymph node dissection around the inferior mesenteric artery with preservation of the left colic artery for rectal cancer.

DETAILED DESCRIPTION:
During surgery for rectal cancer, there is considerable controversy regarding the optimal level of ligation of the inferior mesenteric artery.There has been a differentiation between a high versus low ligation of the inferior mesenteric artery related to whether or not the ligation is above (high ligation) or below (low ligation) the left colic artery. Several studies have demonstrated the benefit of high ligation of the inferior mesenteric artery for the rectal cancer in order to achieve block dissection of lymph node metastases along the root of the inferior mesenteric artery. Excision of the apical lymph node at the root of the inferior mesenteric artery is thought to be necessary for radical resection of rectal cancer because apical lymph node resection contributes to improve lymph node retrieval rates and the accuracy of tumour staging. In contrast, other studies have shown a significant decrease in blood flow after inferior mesenteric artery clamping that may increase the risk of anastomotic ischemia. Patients with high ligation of inferior mesenteric artery had a 3.8 times higher chance of leaking than those with low ligation. Several studies confirmed that the long-term outcomes were not significantly different between high ligation of the inferior mesenteric artery and low ligation. So, a modified procedure was suggested to dissect fatty tissues and nodes in the angle between the inferior mesenteric artery and left colic artery and the artery was ligated below the left colic artery, which represented a compromise between the high and low ligation. Recently, several studies have described laparoscopic lymph node dissection around the inferior mesenteric artery with preservation of the left colic artery for rectosigmoid colon cancer. However, there are a few reports that describe the clinical outcomes associated with this management strategy. Furthermore, the long-term outcomes for laparoscopic lymphadenectomy around the inferior mesenteric artery with rectal cancer have seldom been reported. In the present clinical trial, the investigators perform laparoscopic surgery with this management strategy in rectal cancer. Thus, the goal of this study is to investigate the short-term and oncologic long-term outcomes associated with laparoscopic lymph node dissection around the inferior mesenteric artery with preservation of the left colic artery for rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. pathological confirmed rectal adenocarcinoma
2. solitary radical resectable tumors
3. tumor located at 5-15cm from the anus

Exclusion Criteria:

1. recurrent cases
2. emergency including obstruction, bleeding or perforation
3. severe abdominal adhesions
4. severe malnutrition can not be improved before surgery
5. can not tolerate to surgery due to severe comorbidities of heart, lung, liver or kidney
6. refractory hypoproteinemia or diabetes mellitus
7. previous or concomitant other cancers
8. the patients performed APR or hartmann surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-04; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
anastomotic leak rate | 30 days since the date of surgery
  percentage of patients occuring anastomotic leak within 30 days since surgery
Number of lymph node dissection | 10 days since the date of surgery
Overall survival rate | 3 years since the date of surgery
  3 years total survival rate after surgery
disease-free survival rate | 3 years since the date of surgery
  3 years disease-free survival rate after surgery

SECONDARY OUTCOMES:
30-day mortality rate | within 30 days since the date of surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Tanaka J, Nishikawa T, Tanaka T, Kiyomatsu T, Hata K, Kawai K, Kazama S, Nozawa H, Yamaguchi H, Ishihara S, Sunami E, Kitayama J, Watanabe T. Analysis of anastomotic leakage after rectal surgery: A case-control study. Ann Med Surg (Lond). 2015 May 11;4(2):183-6. doi: 10.1016/j.amsu.2015.05.002. eCollection 2015 Jun. PMID 26042185
- [Result] Cirocchi R, Trastulli S, Farinella E, Desiderio J, Vettoretto N, Parisi A, Boselli C, Noya G. High tie versus low tie of the inferior mesenteric artery in colorectal cancer: a RCT is needed. Surg Oncol. 2012 Sep;21(3):e111-23. doi: 10.1016/j.suronc.2012.04.004. Epub 2012 Jul 6. PMID 22770982
- [Result] Bonnet S, Berger A, Hentati N, Abid B, Chevallier JM, Wind P, Delmas V, Douard R. High tie versus low tie vascular ligation of the inferior mesenteric artery in colorectal cancer surgery: impact on the gain in colon length and implications on the feasibility of anastomoses. Dis Colon Rectum. 2012 May;55(5):515-21. doi: 10.1097/DCR.0b013e318246f1a2. PMID 22513429
- [Result] Cirocchi R, Farinella E, Trastulli S, Desiderio J, Di Rocco G, Covarelli P, Santoro A, Giustozzi G, Redler A, Avenia N, Rulli A, Noya G, Boselli C. High tie versus low tie of the inferior mesenteric artery: a protocol for a systematic review. World J Surg Oncol. 2011 Nov 9;9:147. doi: 10.1186/1477-7819-9-147. PMID 22071020
- [Result] Seike K, Koda K, Saito N, Oda K, Kosugi C, Shimizu K, Miyazaki M. Laser Doppler assessment of the influence of division at the root of the inferior mesenteric artery on anastomotic blood flow in rectosigmoid cancer surgery. Int J Colorectal Dis. 2007 Jun;22(6):689-97. doi: 10.1007/s00384-006-0221-7. Epub 2006 Nov 3. PMID 17082922
- [Result] Trencheva K, Morrissey KP, Wells M, Mancuso CA, Lee SW, Sonoda T, Michelassi F, Charlson ME, Milsom JW. Identifying important predictors for anastomotic leak after colon and rectal resection: prospective study on 616 patients. Ann Surg. 2013 Jan;257(1):108-13. doi: 10.1097/SLA.0b013e318262a6cd. PMID 22968068